CLINICAL TRIAL: NCT03963427
Title: GoBreast - a Prospective Randomized Trial on Breast Reconstruction Methods
Brief Title: Quality of Life, Aesthetic Result and Health Economy in Breast Reconstruction
Acronym: GoBreast
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bröst-07:2-4
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Female; Surgery--Complications
Keywords: breast reconstruction; plastic surgery; microsurgery
MeSH Terms: interventions — Mammaplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Irradiated women (Other): Irradiated women are randomized to reconstruction with a latissimus Dorsi flap and an implant or a deep inferior epigastria perforator flap.
  Interventions: Procedure: Breast reconstruction
- Non-irradiated women (Other): Non-irradiated women are randomized to reconstruction with a thoracodorsal flap with an implant or with an expander and later a permanent implant in two stages.
  Interventions: Procedure: Breast reconstruction

INTERVENTIONS:
Procedure: Breast reconstruction — Irradiated women are randomized to reconstruction with a latissimus Dorsi flap and an implant or a deep inferior epigastria perforator flap. Non-irradiated women are randomized to reconstruction with a thoracodorsal flap with an implant or with an expander and later a permanent implant in two stages.

SUMMARY:
A randomized clinical trial with two arms: irradiated women and non-irradiated women. Irradiated women are randomized to reconstruction with a latissimus Dorsi flap and an implant or a deep inferior epigastria perforator flap. Non-irradiated women are randomized to reconstruction with a thoracodorsal flap with an implant or with an expander and later a permanent implant in two stages.

ELIGIBILITY:
Irradiated patients:

Inclusion Criteria:

* Age 18-60
* DIEP is technically possible
* Unilateral mastectomy
* BMI<30

Exclusion Criteria:

* Scars on abdomen or back
* Bilateral mastectomy
* Previous liposuction abdomen
* 61 years of age or older

Non-irradiated patients

Inclusion Criteria:

->18 years of age

* Unilateral mastectomy
* BMI<30

Exclusion Criteria:

* Bilateral mastectomy
* extensive scars on thorax

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2008-03-08 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Aesthetic outcome | 1 year post-operatively
  Photo evaluations

SECONDARY OUTCOMES:
Breast related quality of life and satisfaction | Pre-operatively and 3 years post-operatively
  Breast-q. Measures breast related quality of life on a scale 1-100. A higher score indicates a higher quality of life.
General quality of life measurement used for health economics | Pre-operatively and 3 years post-operatively
  EuroQol-5 domensions-3 levels is a generic instrument developed for health economic and clinical evaluation of healthcare. A total score between 0 and 1 is calculated. Zero equals death and 1 perfect health.
Depression | Pre-operatively and 3 years post-operatively
  Beck Depression Inventory (BDI 21) for mood assessment. Scale range is 0-63 and higher scores indicate worse outcome.
General quality of life | Pre-operatively and 3 years post-operatively
  Short form health survey (SF-36). The scale ranges from 0 to 100 and a higher score indicates a better quality of life.
Early complication frequency | 2 weeks post-operatively
  Complications described according to Clavien-Dindo
Long-term complications | Five years post-operatively
  Re-operations and corrections
Health economics | Five years post-operatively
  Costs of different procedures
Implant survival (Ancillary study) | 19 years
  Analysis of number of implants removed over time (Ethical permit: 2021-06131-02)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brorson F, Thorarinsson A, Kolby L, Elander A, Hansson E. Early complications in delayed breast reconstruction: A prospective, randomized study comparing different reconstructive methods in radiated and non-radiated patients. Eur J Surg Oncol. 2020 Dec;46(12):2208-2217. doi: 10.1016/j.ejso.2020.07.010. Epub 2020 Jul 26. PMID 32807615
- [Result] Brorson F, Elander A, Thorarinsson A, Hansson E. Patient Reported Outcome and Quality of Life After Delayed Breast Reconstruction - An RCT Comparing Different Reconstructive Methods in Radiated and Non-radiated Patients. Clin Breast Cancer. 2022 Dec;22(8):753-761. doi: 10.1016/j.clbc.2022.09.004. Epub 2022 Sep 17. PMID 36210311
- [Result] Thorarinsson A, Frojd V, Kolby L, Liden M, Elander A, Mark H. Patient determinants as independent risk factors for postoperative complications of breast reconstruction. Gland Surg. 2017 Aug;6(4):355-367. doi: 10.21037/gs.2017.04.04. PMID 28861376
- [Result] Thorarinsson A, Frojd V, Kolby L, Ljungdal J, Taft C, Mark H. Long-Term Health-Related Quality of Life after Breast Reconstruction: Comparing 4 Different Methods of Reconstruction. Plast Reconstr Surg Glob Open. 2017 Jun 21;5(6):e1316. doi: 10.1097/GOX.0000000000001316. eCollection 2017 Jun. PMID 28740762
- [Result] Thorarinsson A, Frojd V, Kolby L, Modin A, Lewin R, Elander A, Mark H. Blood loss and duration of surgery are independent risk factors for complications after breast reconstruction. J Plast Surg Hand Surg. 2017 Oct;51(5):352-357. doi: 10.1080/2000656X.2016.1272462. Epub 2017 Jan 26. PMID 28122466
- [Result] Thorarinsson A, Frojd V, Kolby L, Lewin R, Molinder N, Lundberg J, Elander A, Mark H. A retrospective review of the incidence of various complications in different delayed breast reconstruction methods. J Plast Surg Hand Surg. 2016;50(1):25-34. doi: 10.3109/2000656X.2015.1066683. Epub 2015 Sep 11. PMID 26360138
- See also: Research group — https://www.gu.se/forskning/rekonstruktiv-brostkirurgi